CLINICAL TRIAL: NCT00787982
Title: Pilot Study Evaluating the Feasibility of Real-Time, Magnetic Resonance Thermal Imaging and Magnetic Resonance Imaging-Guided Laser Induced Thermal Therapy for Treatment of Metastatic Brain Tumors
Brief Title: Magnetic Resonance Imaging-Guided Laser Induced Thermal Therapy for Treatment of Metastatic Brain Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Visualase, Inc. (Industry)
Responsible Party: Michael Schulder, MD , Vice Chairman , Department of Neurosurgery, North Shore LIJ Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIS-BR-08-001
Record Dates: First submitted 2008-10-29; First posted 2008-11-10 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Brain Neoplasms
Keywords: brain; metastasis; neoplasm; tumor; Patients with secondary brain neoplasms; laser therapy; laser interstitial thermal therapy
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MRI-Guided Laser Induced Thermal Therapy — LITT uses laser light to heat and destroy the affected tissue; this is sometimes referred to as tissue ablation. In LITT, small fiber-optic applicators are placed directly into the tumor and heating is performed from the inside out, which may lead to the destruction of the tumor

SUMMARY:
In this study, the Visualase Thermal Therapy System will be used on metastatic brain tumors that cannot be removed by surgery. Researchers want to find out if it is possible to use this new device in subjects with 1-3 metastatic brain tumor(s), each measuring 3 centimeters (cm) or smaller. The safety of the device will also be studied.

DETAILED DESCRIPTION:
The Visualase Thermal Therapy System is FDA-cleared for thermal destruction of soft tissue in neurosurgery under MRI guidance. The device combines 3 previously FDA-cleared devices: the Visualase Cooled Laser Application System, which delivers the laser (energy) to the tumor tissue; the PhoTex , Diode Laser Series, which is the laser itself; and the Visualase ENVISION Workstation, which is the computer system that helps the surgeon plan and monitor your treatment.

The Visualase Thermal Therapy System will be used in this study to give subjects a type of therapy called Laser Interstitial Thermal Therapy (LITT). LITT uses laser light to heat and destroy the affected tissue; this is sometimes referred to as tissue ablation. In LITT, small fiber-optic applicators are placed directly into the tumor and heating is performed from the inside out, which may lead to the destruction of the tumor. During the heating process, MRTI can be used to watch the temperatures around the applicator to make sure that the tumor receives enough treatment and that the normal tissues around the tumor do not get too hot.

ELIGIBILITY:
Inclusion Criteria:

* Patient or family able and willing to give informed consent.
* Subjects with metastatic cancer to the brain who have failed at least one conventional therapy (surgery, stereotactic radiosurgery, and/or whole brain radiotherapy).
* Three or fewer previously treated or untreated lesion(s) in the brain.
* Tumor size ≤ 3.0 cm in largest diameter.
* MR imaging is not contraindicated for the patient.
* Lesion(s) are clearly defined on pre-therapy contrast enhanced MRI scans as determined by the treating surgeon.
* Able and willing to attend all study visits.
* Karnofsky Performance Scale score >70 for patients over the age of 15.
* Lansky Play Scale >70 for patients 15 years of age or younger.

Exclusion Criteria:

* Patients or family unwilling or unable to give written consent.
* Patients who cannot physically fit in, or are too heavy for, the MRI scanner.
* Patients with contra-indications to MRI imaging, such as, but not limited to, pacemakers or defibrillators, non-compatible aneurysm clips, shrapnel, or other internal ferromagnetic objects.
* Known sensitivity to gadolinium-DTPA.
* Based on Treatment Planning Imaging (MR and/or CT):

  * Brain edema and/or mass effect that causes midline shift or shift in wall of ventricle of more than 5 mm.
  * Lesions localized in the brain stem.
  * Lesions less than 5mm from primary branches of cerebral vessels, venous sinus, hypophysis or cranial nerves.
  * Evidence of recent (<2 weeks) hemorrhage.
* Presence of more than 3 brain tumors at the time of enrollment.
* Symptoms and signs of increased intracranial pressure.
* Medical issues which prohibit the patient from undergoing surgery (as determined by the treating surgeon, anesthesiologist, IMPAC clinic, referring physician).
* Patients who are unable to receive corticosteroids.
* Positive pregnancy test for women of child-bearing age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Rate of technical success or failure to complete the initial procedure with no associated major complications. | within 24 hours following the procedure

SECONDARY OUTCOMES:
Examination of the extent to which Visualase predictions based on MRTI data match lesion dimensions form post-therapy MRI assessments. | Immediately following treatment (day 0)
Estimates of durations, required facilities, required personnel, and costs for all aspects of the treatment procedure | from day 0 to patient release
Local control of treated lesions as defined by volume of lesions increasing by no more than 25% | Day 30, 90, and 180 days post procedure
Accrual of patient survival post Visualase therapy | Sooner of 3 years or patient death
Procedure-related morbidity and mortality | 30, 90,180 days post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

REFERENCES:
- See also: Sponsors website — http://www.visualaseinc.com